CLINICAL TRIAL: NCT03778034
Title: Effect of Forward Head Posture(FHP) on Temopromandibular Joint (TMJ) Proprioception in Post-pubertal Females
Brief Title: Effect of Forward Head Posture(FHP)on Temopromandibular Joint (TMJ) Proprioception in Post-pubertal Females
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HAhmed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, HAhmed, lecturer at biomechanics department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/001886
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female with forward head posture: post-pubertal females suffering from (FHP) with Craniovertebral angle (CVA) less than 49 degrees(study group)
  Interventions: Other: female with Forward head posture
- healthy female without (FHP): post-pubertal females expected to exhibit an average normal CVA within 10degrees range from 49 to 59 (control group)
  Interventions: Other: healthy female without (FHP)

INTERVENTIONS:
Other: female with Forward head posture — measuring tmj proprioception with open eyes and closed eyes for mouth opening,right deviation,left deviation and protrusion,cranio vertebral angle and shoulder angle
  Groups: Female with forward head posture
Other: healthy female without (FHP) — measuring tmj proprioception with open eyes and closed eyes for mouth opening,right deviation,left deviation and protrusion,cranio vertebral angle and shoulder angle
  Groups: healthy female without (FHP)

SUMMARY:
No studies up to date has been evaluated the effect of FHP on TMJ proprioception.Therefore, this study will be the first one which aims to investigate the effect of FHP on TMJ proprioception in post-pubertal females

DETAILED DESCRIPTION:
Forward head posture and temporomandibular disorder are two common problems in post-pubertal females. They are closely related to each other. Previous studies showed influences of head posture on the mandibular rest position, range of functional movements and the jaw and neck muscles work together during rhythmic movements. They affirm that patients with TMD present more alterations in head positioning than patients with no dysfunction .

However, no studies up to date has been evaluated the effect of FHP on TMJ proprioception. The proprioceptors in the human TMJ play important key role in identification of mandibular position when the teeth are not occluded. TMJ receptors provide the greater afferent activity regarding perceptual awareness of joint position and movement . Proper assessment of TMJ proprioception may be critical for designing not only rehabilitation but also pre-habilitation interventions for patients with FHP aiming to prevent TMD. Therefore, this study will be the first one which aims to investigate the effect of FHP on TMJ proprioception in post-pubertal females. This study may expand the role of physiotherapy in woman's health.

ELIGIBILITY:
Inclusion Criteria:

1. They should be at least 1 year post-puberty.
2. Their age will range from 14 to 19 years old.
3. Their body mass index (BMI) will range from 18-25 kg/m2.
4. They should spend long period of time with bad posture on computer, laptop or smart phones.

Exclusion Criteria:

* They shouldn't have headache, migraine, vertebra-basilar insufficiency,temporo mandibular disorders (TMD) ,uncorrected impairment of vision or audition, neck pain, fixed or mobile spinal deformity or history of fracture or surgery of the upper quadrant of the body

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Forward head posture and temporomandibular disorder are two common problems in post-pubertal females.Females exhibit more incidence of FHP after puberty than males. This posture of greater flexion in females can be attributable to psychosocial issues, such as stress, or partly associated with the development of secondary sex characteristics in females.Temporomandibular disorders (TMD) are common pain conditions that have the highest prevalence among females of reproductive age.the male to female ratio of TMD patients is estimated at around 1:3 and The pattern of onset after puberty and lowered prevalence rates in the postmenopausal years suggest that female reproductive hormones may play an etiologic role in TMD
Study Population: Proper assessment of TMJ proprioception may be critical for designing not only rehabilitation but also pre-habilitation interventions for patients with FHP aiming to prevent TMD. Therefore, this study will be the first one which aims to investigate the effect of FHP on TMJ proprioception in post-pubertal females. This study may expand the role of physiotherapy in woman's health.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-11-10 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Testing TMJ proprioception | one month
  TMJ proprioception will be tested through a digital vernier caliper for each female in both groups. Each female will be asked to sit on a stool, feet will be rested on the floor, arms will be supported on armrests, knees and elbow joints will assume right angles, and the chair's back will not exceed suprascapular border. With closed eyes, the female's mouth will be opened passively by 3 cm measured by adigital Vernier caliper, which is considered as functional position of jaw for eating and speech. The procedures will be repeated 3 times and maintained for 3 seconds. Then, each female will be asked to open her mouth actively for the target distance and the distance will bemeasured by the caliper.

SECONDARY OUTCOMES:
measuring the shoulder angle | one month
  The angle formed at the intersection of the line between the midpoint of the humerus and spinous process of C7 and the horizontal line through the midpoint of the humerus. The investigators considered 52° as the reference angle and will be measure like CVA

CONTACTS AND LOCATIONS:
Overall Officials: amel youssef, phd, Principal Investigator — Cairo University